CLINICAL TRIAL: NCT00092092
Title: A Double-Blind, Double-Dummy, Randomized, Placebo-Controlled, 2-Arm, 2X2 Crossover Study Comparing the Effects of Montelukast, Inhaled Budesonide, and Placebo on Lower Leg Growth in Children (Prepubertal, Tanner Stage I) With Mild Asthma
Brief Title: Study of Montelukast and Its Effect on Lower Leg Growth in Children With Asthma (MK-0476-254)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0476-254; 2004_023 (Other: Telerx ID Number)
Record Dates: First submitted 2004-09-21; First posted 2004-09-24 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2022-02

CONDITIONS: Asthma, Bronchial
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Montelukast→Placebo (Experimental): Participants receive one montelukast 5 mg chewable tablet once daily (QD) for 3 weeks. After a 2-week washout period, participants receive one placebo chewable tablet QD for 3 weeks.
  Interventions: Drug: Montelukast chewable tablets; Drug: Placebo to montelukast chewable tablets
- Placebo→Montelukast (Experimental): Participants receive one placebo chewable tablet QD for 3 weeks. After a 2-week washout period, participants receive one montelukast 5 mg chewable tablet QD for 3 weeks.
  Interventions: Drug: Montelukast chewable tablets; Drug: Placebo to montelukast chewable tablets
- Budesonide→Placebo (Active Comparator): Participants receive budesonide 200 mcg inhalation powder twice daily (BID) for 3 weeks. After a 2-week washout period, participants receive placebo inhalation powder BID for 3 weeks.
  Interventions: Drug: Budesonide inhaler; Drug: Placebo to budesonide inhaler
- Placebo→Budesonide (Active Comparator): Participants receive placebo inhalation powder BID for 3 weeks. After a 2-week washout period, participants receive budesonide 200 mcg inhalation powder BID for 3 weeks.
  Interventions: Drug: Budesonide inhaler; Drug: Placebo to budesonide inhaler

INTERVENTIONS:
Drug: Montelukast chewable tablets — Montelukast sodium 5 mg chewable tablets
  Arms: Montelukast→Placebo; Placebo→Montelukast
Drug: Budesonide inhaler — Budesonide 200 mcg inhalation powder
  Arms: Budesonide→Placebo; Placebo→Budesonide
Drug: Placebo to montelukast chewable tablets — Placebo chewable tablets
  Arms: Montelukast→Placebo; Placebo→Montelukast
Drug: Placebo to budesonide inhaler — Placebo inhalation powder
  Arms: Budesonide→Placebo; Placebo→Budesonide

SUMMARY:
The purpose of this study is to determine the effect of montelukast, an approved medication, on the lower leg growth rate in children with mild asthma. The primary hypothesis is that the lower leg length (LLL) growth rate for children treated with montelukast compared to placebo will be established.

DETAILED DESCRIPTION:
This is a crossover study that consists of a 2-week placebo run-in period, then a first 3-week treatment period, then a 2-week washout period, and then a second 3-week treatment period. Participants will be randomized to treatment with either montelukast and placebo or budesonide and placebo. The duration of treatment is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A 6-month history of asthma with periodic episodes requiring treatment.

Exclusion Criteria:

* Medical history of a lung disorder (other than asthma) or a recent upper respiratory tract infection.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2002-10; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Short-term lower-leg growth rate (LLGR) | Baseline and Week 3
  Lower leg length was measured in millimeters (mm) using a knemometer.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Pedersen S, Agertoft L, Williams-Herman D, Kuznetsova O, Reiss TF, Knorr B, Dass SB, Wolthers OD. Placebo-controlled study of montelukast and budesonide on short-term growth in prepubertal asthmatic children. Pediatr Pulmonol. 2007 Sep;42(9):838-43. doi: 10.1002/ppul.20666. PMID 17659605